CLINICAL TRIAL: NCT04771117
Title: Defiances to Face COVID-19 Pandemic in Mexico
Status: Completed | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, GONZALEZ-OJEDA ALEJANDRO, Principal Investigator, Instituto Mexicano del Seguro Social
Other Study IDs: Fear5
Record Dates: First submitted 2021-02-03; First posted 2021-02-25 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Health Behavior; Risk-Taking; Covid19
Keywords: Health Behavior; Pandemic; Risk-Taking; Mexico; Covid-19
MeSH Terms: conditions — Health Behavior; Risk-Taking; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Fear of Covid-19 Scale — The Fear of Covid-19 Scale (FCV-19S) is a questionnaire that evaluates fear of the global pandemic caused by the SARS-CoV-2. The FVC-19S consists of seven items, such as "It makes me uncomfortable to think about coronavirus-19," "I am afraid of losing my life because of coronavirus-19," and "When watching news and stories about coronavirus-19 on social media, I become nervous or anxious," each with a five-point Likert scale of options. The participant is instructed to choose the option that best represents their perception about the statement presented. The maximum possible total is 35 points. The scale's authors indicate that the higher the score is, the higher is the level of the participants' fear of COVID-19.

SUMMARY:
The aim of this study is to identify the risk factors favoring the contagion of COVID-19 by studying the quarantine behavior and preventive measures in the Mexican population. As a secondary aim, the investigators sought to identify areas that need reinforcement, to help develop strategies for a successful plan to face an upcoming pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Being Mexican or residents of the country
* Participants over 15 years

Exclusion Criteria:

* Participants under 15 years of age
* Participants with incomplete surveys
* Being a tourist currently staying in the country or being Mexican residing in another country

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study sample was the Mexican general population currently living in the covid-19 pandemic.
Sampling Method: Non-Probability Sample
Enrollment: 4004 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Risk Factors | Baseline
  Risk factors favoring the contagion of COVID-19 by studying the quarantine behavior and preventive measures in the Mexican population.

SECONDARY OUTCOMES:
Fear of Covid-19 | Baseline
  The Fear of Covid-19 Scale (FCV-19S) is a questionnaire that evaluates fear of the global pandemic caused by the SARS-CoV-2. The FVC-19S consists of seven items, such as "It makes me uncomfortable to think about coronavirus-19," "I am afraid of losing my life because of coronavirus-19," and "When watching news and stories about coronavirus-19 on social media, I become nervous or anxious," each with a five-point Likert scale of options. The participant is instructed to choose the option that best represents their perception about the statement presented. The maximum possible total is 35 points. The scale's authors indicate that the higher the score is, the higher is the level of the participants' fear of COVID-19.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Mexicano del Seguro Social, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Derived] Ibarrola-Pena JC, Barbosa-Camacho FJ, Almanza-Mena YL, Chejfec-Ciociano JM, Reyes-Elizalde EA, Romero-Limon OM, Zaragoza-Organista R, Cervantes-Perez E, Sapien-Fernandez JH, Guzman-Barba JA, Flores-Becerril P, Ochoa-Rodriguez I, Najar-Hinojosa R, Cueto-Valadez AE, Cueto-Valadez TA, Lopez-Zendejas M, Fuentes-Orozco C, Cervantes-Guevara G, Miranda-Ackerman RC, Gonzalez-Ojeda A. Preventive measures against the COVID-19 pandemic in Mexico: A cross-sectional study. Front Public Health. 2022 Oct 11;10:932010. doi: 10.3389/fpubh.2022.932010. eCollection 2022. PMID 36304240